CLINICAL TRIAL: NCT06699212
Title: A Phase 3 Multicenter, Randomized, Open-label Study of ASP-1929 Photoimmunotherapy in Combination With Pembrolizumab Versus Standard of Care in the First-line Treatment of Patients With Locoregional Recurrence of Squamous Cell Carcinoma of the Head and Neck (HNSCC) With No Distant Metastases
Brief Title: A Study of ASP-1929 Photoimmunotherapy in Combination With Pembrolizumab in First-line Treatment of Locoregional Recurrent Squamous Cell Carcinoma of the Head and Neck With No Distant Metastases
Acronym: ECLIPSE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Rakuten Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP-1929-381; ECLIPSE (Other: Rakuten Medical)
Record Dates: First submitted 2024-08-07; First posted 2024-11-21 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma
Keywords: HNSCC; Squamous Cell Carcinoma of Head and Neck; Head and Neck Squamous Cell Carcinoma; Oral Cavity Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Head and Neck; immunotherapy; medical device; laser phototherapy; Epidermal Growth Factor Receptor; PD-1 Inhibitor; Immune Checkpoint Inhibitor; Alluminox; Rakuten Medical; ASP-1929; photoimmunotherapy; head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab; Carboplatin; Cisplatin; Fluorouracil; Paclitaxel; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- 320 mg/m^2 ASP-1929 Photoimmunotherapy + pembrolizumab (Experimental): ASP-1929 320 mg/m^2 IV infusion followed by illumination with 690 nm red light at accessible tumor sites using the investigational PIT690 Laser System (24 ± 4 hours after end of ASP-1929 infusion). Treatment with ASP-1929 PIT will be repeated every 4 to 6 weeks depending on clinical judgement of investigators.
  Pembrolizumab: 200 mg every 3 weeks (Q3W) IV infusion over 30 minutes for the first 6 cycles. After the first 6 cycles, pembrolizumab dosing regimen can be converted from 200 mg Q3W to 400 mg every 6 weeks (Q6W) at the investigator's discretion.
  Treatment in the experimental arm will start with the infusion of pembrolizumab on Cycle 1 Day 1 (C1D1) after which ASP-1929 Photoimmunotherapy will follow 7 days later, on Treatment 1 Day 1 (T1D1). Patients will be treated with ASP-1929 PIT and pembrolizumab for up to 24 months.
  Interventions: Combination Product: ASP-1929 Photoimmunotherapy; Biological: Pembrolizumab
- 640 mg/m^2 ASP-1929 Photoimmunotherapy + pembrolizumab (Experimental): ASP-1929 640 mg/m^2 IV infusion followed by illumination with 690 nm red light at accessible tumor sites using the investigational PIT690 Laser System (24 ± 4 hours after end of ASP-1929 infusion). Treatment with ASP-1929 PIT will be repeated every 4 to 6 weeks depending on clinical judgement of investigators.
  Pembrolizumab: 200 mg every 3 weeks (Q3W) IV infusion over 30 minutes for the first 6 cycles. After the first 6 cycles, pembrolizumab dosing regimen can be converted from 200 mg Q3W to 400 mg every 6 weeks (Q6W) at the investigator's discretion.
  Treatment in the experimental arm will start with the infusion of pembrolizumab on Cycle 1 Day 1 (C1D1) after which ASP-1929 Photoimmunotherapy will follow 7 days later, on Treatment 1 Day 1 (T1D1). Patients will be treated with ASP-1929 PIT and pembrolizumab for up to 24 months.
  Interventions: Combination Product: ASP-1929 Photoimmunotherapy; Biological: Pembrolizumab
- Pembrolizumab or pembrolizumab + chemotherapy (Control) (Active Comparator): Patients in the control arm will receive physician's choice SOC. Patients randomized to SOC may only be treated with one of the following SOC options:
  1. Pembrolizumab alone
  2. Pembrolizumab + platinum (cisplatin or carboplatin) + 5-fluorouracil (5-FU) or taxane (paclitaxel or docetaxel)
  Pembrolizumab: 200 mg Q3W IV infusion over 30 minutes for the first 6 cycles. After the first 6 cycles, pembrolizumab administration can be switched from 200 mg Q3W to 400 mg Q6W at the investigator's discretion.
  Cisplatin or carboplatin: AUC 5 mg/mL/min or 100 mg/m^2 IV infusion on Day 1 of each cycle, Q3W for up to 6 cycles
  5-FU: 1000 mg/m^2 IV infusion per day from Days 1-4 of each cycle, Q3W for up to 6 cycles
  Paclitaxel: At investigator's choice, 100 mg/m^2 IV infusion on Day 1 and Day 8 of each 21-day cycle or paclitaxel 175 mg/m^2 IV infusion on Day 1 of each 21-day cycle for up to 6 cycles
  Docetaxel: 75 mg/m^2 IV infusion on Day 1 of each cycle, Q3W for up to 6 cycles
  Interventions: Biological: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: 5-fluorouracil; Drug: Paclitaxel; Drug: Docetaxel

INTERVENTIONS:
Combination Product: ASP-1929 Photoimmunotherapy — ASP-1929 IV infusion followed by illumination with light dose of 50 J/cm^2 for superficial lesions and 100 J/cm for interstitial lesions within 24 +/- 4 hours after the end of ASP-1929 infusion (up to 24 months)
  Other Names: cetuximab sarotalocan; PIT690 Laser System
  Arms: 320 mg/m^2 ASP-1929 Photoimmunotherapy + pembrolizumab; 640 mg/m^2 ASP-1929 Photoimmunotherapy + pembrolizumab
Biological: Pembrolizumab — 200 mg Q3W or 400 mg Q6W, IV infusion over 30 minutes (up to 24 months)
  Other Names: Keytruda
Drug: Carboplatin — Area under the curve (AUC) 5 mg/mL/min IV infusion, Q3W up to 6 cycles
  Arms: Pembrolizumab or pembrolizumab + chemotherapy (Control)
Drug: Cisplatin — 100 mg/m^2 IV infusion, Q3W up to 6 cycles
  Arms: Pembrolizumab or pembrolizumab + chemotherapy (Control)
Drug: 5-fluorouracil — 1000 mg/m^2 per day from Days 1-4 of each cycle, IV infusion, Q3W up to 6 cycles
  Arms: Pembrolizumab or pembrolizumab + chemotherapy (Control)
Drug: Paclitaxel — 100 mg/m^2 IV infusion given on Days 1 and 8, Q3W up to 6 cycles or 175 mg/m^2 IV infusion given on Day 1, Q3W up to 6 cycles
  Arms: Pembrolizumab or pembrolizumab + chemotherapy (Control)
Drug: Docetaxel — 75 mg/m^2 IV Infusion, Q3W up to 6 cycles
  Arms: Pembrolizumab or pembrolizumab + chemotherapy (Control)

SUMMARY:
The goal of this clinical trial is to learn if ASP-1929 photoimmunotherapy (PIT) in combination with pembrolizumab works to treat recurrent squamous cell cancer of the head and neck (HNSCC) with no distant metastases. It will also learn about the safety of ASP-1929 PIT in combination with pembrolizumab.

Researchers will compare ASP-1929 PIT in combination with pembrolizumab to pembrolizumab alone or pembrolizumab plus chemotherapy (carboplatin or cisplatin, plus 5-fluorouracil or paclitaxel or docetaxel) according to physician's choice (control arm).

The overall primary study hypothesis being tested is whether ASP-1929 PIT plus pembrolizumab combination treatment improves the overall survival (OS) of the population defined by the inclusion/exclusion criteria over the control arm.

DETAILED DESCRIPTION:
This is a phase 3 multicenter, randomized study designed to evaluate the efficacy and safety of ASP-1929 photoimmunotherapy (PIT) in combination with pembrolizumab versus pembrolizumab-based standard of care (SOC) as first-line treatment of locoregional recurrent HNSCC in patients with no distant metastases.

Patients will be enrolled into the study starting with 3 treatment arms, ASP-1929 PIT at doses of 320 mg/m^2 or 640 mg/m^2 in combination with pembrolizumab treatment arms or a SOC treatment arm in which patients may receive pembrolizumab alone or pembrolizumab plus chemotherapy according to physician's choice.

Treatment assignment within the SOC treatment arm will be based on the decision of the site investigator. To ensure that the SOC treatment arm is appropriately balanced, a 50% enrollment cap will be imposed on pembrolizumab monotherapy and pembrolizumab plus chemotherapy, so that approximately the same number of patients will have been treated within each category.

At the start of the study all patients will be randomized 2:2:1 ratio to ASP-1929 PIT 320 mg/m^2 plus pembrolizumab versus ASP-1929 PIT 640 mg/m^2 plus pembrolizumab versus SOC (pembrolizumab alone or pembrolizumab plus chemotherapy according to physician's choice).

An interim analysis (IA) will be conducted for this study as part of the dose optimization process. Patient enrollment will continue during the period of preparation and conduct of this IA. Based on the findings from the first interim analysis (IA1), the Sponsor will have the option to close one of the two ASP-1929 PIT treatment arms for enrollment. The final decision on the optimized ASP-1929 PIT dose for this study will be made in agreement with the US Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological evidence of squamous cell carcinoma of a head and neck primary site (per American Joint Committee on Cancer [AJCC], other than nasopharynx or cuSCC).
* Appropriate for SOC first-line treatment of their recurrent head and neck cancer with pembrolizumab ± chemotherapy.
* No known history of any distant metastatic disease (M1 by AJCC eighth edition).
* Tumors with at least one PIT-accessible and RECIST 1.1 measurable lesion as assessed by investigator.
* Anti-PD-1 and anti-PD-L1-treatment naïve.
* Combined positive score (CPS) ≥ 1 as determined locally by an FDA-approved test
* Have results from testing of human papillomavirus (HPV) status for oropharyngeal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at the time of screening
* Adequate hematologic, renal, and hepatic organ function
* Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening and must be willing to use a highly effective birth control while on study or be surgically sterile or abstain from heterosexual sexual activity for the course of the study through 180 days after the last dose of study treatment. Male patients must agree to use a highly effective method of contraception starting with the first dose of study medication through 120 days after the last dose of study treatment.

Exclusion Criteria:

* Diagnosed and/or treated for additional malignancy within 2 years before randomization except for those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, basal cell skin cancer, localized prostate cancer, or ductal carcinoma in situ). Patients with a history of other prior cancer treated with complete surgical resection and with no evidence of disease may be eligible based on discussion with the Medical Monitor.
* History of significant (Grade ≥ 3) cetuximab infusion reactions
* Prior allogeneic tissue/solid organ transplant
* Known or active central nervous system metastases and/or carcinomatous meningitis
* Life expectancy of less than 3 months
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Evidence of interstitial lung disease or current active, noninfectious pneumonitis
* Active infection requiring systemic therapies such as antibiotic, antifungal, or antiviral intervention
* Known or active bacterial, viral, or fungal infection including tuberculosis, Hepatitis B (e.g., HBV DNA is detected), or Hepatitis C (e.g., RNA [qualitative] is detected)
* Known history of testing positive for human immunodeficiency virus or acquired immunodeficiency syndrome (AIDS)-related illness
* Prior or ongoing Grade ≥ 3 tumor hemorrhage within 12 weeks of randomization
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior systemic chemotherapy or targeted small molecule therapy or radiation therapy within 2 weeks of C1D1 or has not recovered (i.e., Grade ≤ 1 or at baseline) from adverse events (AEs) due to previously administered agent
* Prior anticancer monoclonal antibody therapy or investigational agent or intervention within 4 weeks of C1D1 or has not recovered (i.e., Grade ≤ 1 or at baseline) from AEs due to previously administered agent
* Prior receipt of ASP-1929 at any time
* Receiving chronic systemic steroid therapy (in doses exceeding 10 mg per day of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to randomization
* Received a live vaccine within 4 weeks of randomization; seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed
* Requiring future examinations or treatments within 4 weeks after an ASP-1929 PIT treatment exposing the patient to significant light (e.g., eye examinations, surgical procedures, endoscopy) that is unrelated to the ASP-1929 PIT treatment
* Major surgery or significant traumatic injury within 4 weeks before randomization, or anticipation of the need for major surgery during the course of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2024-12-24 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to approximately 48 months
  OS is defined as the time from randomization until death due to any cause.

SECONDARY OUTCOMES:
Complete response rate (CRR) per modified Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) as assessed by central reviewer | Up to approximately 48 months
  CRR is defined as the proportion of patients with best overall response of confirmed CR
Overall response rate (ORR) per modified RECIST 1.1 as assessed by central reviewer | Up to approximately 48 months
  ORR is defined as the proportion of patients with best overall response of confirmed CR or confirmed partial response (PR)
Progression-free survival (PFS) per modified RECIST 1.1 as assessed by central reviewer | Up to approximately 48 months
  PFS is defined as the time from randomization to the first documented tumor progression or death due to any cause, whichever occurs first.
OS rates at 12, 18, and 24 months | 12, 18, and 24 months
  OS rates at 12, 18, and 24 months are defined as the proportions of patients who are alive at these time points
Duration of Response (DOR) per modified RECIST 1.1 as assessed by central reviewer | Up to approximately 48 months
  DOR is defined as the time from first response (CR or PR) that is subsequently confirmed to the time of disease progression or death due to any cause, whichever occurs first
Duration of CR per modified RECIST 1.1 as assessed by central reviewer | Up to approximately 48 months
  Duration of CR is defined as the time from first response (CR) that is subsequently confirmed to the time of disease progression or death due to any cause, whichever occurs first
Time to response (TTR) | Up to approximately 25 months
  TTR is defined as the time from randomization to the first confirmed response (CR or PR)
CRR from randomization to End of Treatment as assessed by the central reviewer | Up to approximately 25 months
  CRR (confirmed response) from randomization to end of treatment is defined as the proportion of patients with the best overall response of CR, where the CR occurs anytime during the study treatment period (e.g., CR after Progressive Disease [PD] will be counted).
Proportion of treatment-emergent adverse events (TEAEs) by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | Up to approximately 48 months
  TEAEs refer to any AEs that begin or worsen on or after the start of any study treatment through 30 days after the last dose of study treatment and any additional immune-related adverse events (irAEs) that begin between 30 days and 90 days after the last dose of anti-PD1 treatment. In addition, any serious AE with an onset date more than 30 days after the last dose of study treatment assessed by the investigator as related to study treatment will be considered a TEAE.
Proportion of treatment-related adverse events (TRAEs) by CTCAE v5.0 | Up to approximately 48 months
  Any TEAE (defined in Outcome 10) for which there is a reasonable possibility that the investigational treatment caused the adverse event.
Proportion of serious adverse events (SAEs) by CTCAE v5.0 | Up to approximately 48 months
  An AE or suspected adverse reaction is considered 'serious' if, in the view of either the Investigator or Sponsor, it meets one or more of the following criteria (21 CFR 312.32 (a)): Results in death, Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization, Results in persistent or significant disability/incapacity, or Is a congenital anomaly/birth defect or Important medical event.
Quality of Life assessment: EORTC Core Quality of Life Questionnaire- Core 30 (EORTC QLQ-C30) | Up to approximately 28 months
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Each scale or item score is standardized to a range of 0 to 100. Higher scores on the functional scales reflect better functioning, whereas higher scores on the symptom scales indicate more severe symptoms or greater levels of distress. Similarly, higher scores on the global health status scale denote better overall health and quality of life. Thus, an optimal quality of life profile is characterized by high scores on the functional and global health status scales, combined with low scores on the symptom scales. The summed scores of Functional scales, Symptom scales, and Global health status domains of EORTC-QLQ-C30 are compared between treatment arms.
Quality of Life assessment: EORTC Quality of Life Questionnaire Head and Neck Module (QLQ-H&N35) | Up to approximately 28 months
  EORTC QLQ-H&N35 is a 35-item questionnaire developed to assess QoL of head and neck cancer participants and consists of 7 multi-item scales that assess pain, swallowing, senses, speech, social eating, social contact and sexuality. Each scale or item score is standardized to a range of 0 to 100. Lower score on each scale represents fewer symptoms and less impact on the patient's daily life. The summed scores of the scales of EORTC-QLQ-H&N35 are compared between treatment arms.
Population pharmacokinetics (PK) - Clearance (Experimental Arm Only) | Before the start of 1st ASP-1929 infusion, 0.25 hours, 4 hours, 24 hours, 192 hours, 360 hours after end of 1st infusion; same timepoints for 2nd ASP-1929 infusion
  A structural compartment model with population factors such as age, race, ECOG, and sex will be utilized to analyze concentration levels. The clearance estimates associated with different factors will be reported.
Presence of anti-drug antibodies (ADAs) (Experimental Arm Only) | Before the start of 1st ASP-1929 infusion, 15 days after end of 1st infusion; same timepoints for 2nd ASP-1929 infusion
  Average concentration level of ADAs at baseline and 15 days after ASP-1929 infusion for the first 2 treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Ethan Chen, MD, Study Director — Rakuten Medical, Inc.; Rebecca Cheng, MD, Study Director — Rakuten Medical, Inc.
Locations (22):
- United States (8):
  - City of Hope, Duarte, California
  - University of Miami, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Japan (5):
  - Aichi Cancer Center, Aichi
  - Hiroshima University Hospital, Hiroshima
  - Kyoto Prefectural University of Medicine, Kyoto
  - Tokyo Medical University Hospital, Tokyo
  - Tottori University Hospital, Yonago
- Taiwan (9):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan

IPD SHARING:
Plan to Share IPD: No